CLINICAL TRIAL: NCT05900804
Title: The Effect of Training Prepared in Line With the Fracture Liaison Service Model in Patients Undergoing Hip Surgery on Patients' Fragility Level, Care Dependence, and Fear of Movement: A Randomized Controlled Study
Brief Title: The Effect of Training Prepared in Line With Fracture Liaison Service Model on Frailty in Hip Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Halise Cinar, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Halise03
Record Dates: First submitted 2023-04-16; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Geriatric Patients
Keywords: Nursing; Frailty; Education; Fracture Liaison Services
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): * On the 3rd postoperative day, patient information form, patient follow-up form, Edmonton frailty scale, kinesiophobia causes scale and care dependency scale will be applied in the patient room. Afterwards, the training prepared in line with the fracture liaison service model will be verbally explained to the patients and then the booklet prepared by taking expert opinion will be given to the patients.
  * 3rd week patient follow-up form, Edmonton frailty scale, kinesiophobia causes scale and care dependency scale will be applied in orthopedics and traumatology outpatient clinic.
  * 3rd month patient follow-up form, Edmonton frailty scale, kinesiophobia causes scale and care dependency scale will be applied at home visit.
  Interventions: Other: Training Prepared in Line with the Fracture Liaison Service Model
- Control group (No Intervention): * On the 3rd postoperative day, patient information form, patient follow-up form, Edmonton frailty scale, kinesiophobia causes scale and care dependency scale will be applied in the patient room.
  * Week 3 patient follow-up form, Edmonton frailty scale, kinesiophobia causes scale and care dependency scale will be applied in orthopedics and traumatology outpatient clinic.
  * 3rd month patient follow-up form, Edmonton frailty scale, kinesiophobia causes scale and care dependency scale will be applied at home visit. Afterwards, the training prepared in line with the fracture liaison service model will be verbally explained to the patients and then the booklet prepared by taking expert opinion will be given to the patients.

INTERVENTIONS:
Other: Training Prepared in Line with the Fracture Liaison Service Model — The Effect of Education Prepared in Line with Fracture Liaison Service Model on Patients' Frailty Level, Care Dependency and Fear of Movement in Hip Surgery Patients
  Arms: Intervention Group

SUMMARY:
This study is a randomized controlled experimental research with pretest-posttest control group. The aim of this study is to evaluate the effect of the training prepared in line with the fracture liaison service model on the level of frailty, care dependency and fear of movement in patients undergoing hip surgery. The main questions it aims to answer are as follows:

* Does the training provided to patients undergoing hip surgery in line with the fracture liaison service model have an effect on the level of frailty of patients?
* Does the training provided to patients undergoing hip surgery in line with the fracture liaison service model have an effect on patients' care dependency?
* Does the education given to patients undergoing hip surgery in line with the fracture liaison service model have an effect on patients' fear of movement? It is very important to prevent secondary fractures that may occur in patients undergoing hip surgery. Therefore, the most appropriate prevention interventions to reduce fractures in patients depend on the risk profile and the place of education for hospitalized patients is very important. In this study, Personal Information Collection Form, Patient Follow-up Form, Edmonton Frailty Scale, Causes of Kinesiophobia Scale and Care Dependency Scale will be applied to control and intervention group patients. It is planned to provide training to the intervention group patients in line with the fracture liaison service model. This study will evaluate the effect of the training on patients' level of frailty, care dependency and fear of movement.

DETAILED DESCRIPTION:
The frail patient is a more complex patient group that is difficult for healthcare professionals to monitor and treat. These patients are more prone to undesirable outcomes such as hospitalization and death. The risk of frailty increases even more in the elderly population who experience more health problems, especially in the later stages of old age. In the care of the frail elderly, the nurse, together with the healthcare team, should be able to detect the complications that may develop in the elderly at an early stage, take the necessary precautions and provide services according to the needs. With the education given in line with the risk factors that occur in frail patients, individuals will be informed about frailty, and at the same time, environmental arrangements, exercises, etc. It is thought that the immobilization of the patient and the occurrence of secondary fractures will be minimized with such activities. In order to minimize or prevent possible postoperative complications and to prevent falls and secondary fractures; this study was planned to evaluate the effect of the training prepared in line with the fracture liaison service model on the level of frailty, care dependency and fear of movement in patients undergoing hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Being diagnosed with osteoporosis
* Being conscious and able to answer questions
* Not having a problem that would prevent communication

Exclusion Criteria:

* Under 65 years of age with fractures
* Patients with Parkinson's disease
* Patients with visual and hearing impairment
* Patients undergoing hip surgery for the second time

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Personal Information Collection Form | Baseline
  The form prepared by the researchers with the support of the literature includes questions about the sociodemographic characteristics of the patients (gender, age, height, weight, educational status, etc.). This form will be used in the first interview with the patients.
Patient Follow-up Form | 3 days after the operation
  With this form, complications and problems that patients may experience in the postoperative period will be evaluated and the observed complications and problems will be marked on the patient follow-up form. Patients will be followed up for 3 months with this form
Patient Follow-up Form | 3 weeks after the operation
  With this form, complications and problems that patients may experience in the postoperative period will be evaluated and the observed complications and problems will be marked on the patient follow-up form. Patients will be followed up for 3 months with this form
Patient Follow-up Form | 3 months after the operation
  With this form, complications and problems that patients may experience in the postoperative period will be evaluated and the observed complications and problems will be marked on the patient follow-up form. Patients will be followed up for 3 months with this form
Edmonton Frailty Scale | 3 days after the operation
  Edmonton Frailty Scale was developed by Rolfson et al. (2006) to assess frailty in elderly individuals. The scale consists of 9 frailty dimensions included in the Comprehensive Geriatric Assessment and accepted as determinants of frailty. These frailty dimensions include cognitive status, general health status, functional independence, social support, medication use, nutrition, mood, continence and functional status. The scale consists of 11 items in total. The 'clock test' is used to assess cognitive status and the 'Timed Up and Go test' is used to assess functional performance.
Edmonton Frailty Scale | 3 weeks after the operation
  Edmonton Frailty Scale was developed by Rolfson et al. (2006) to assess frailty in elderly individuals. The scale consists of 9 frailty dimensions included in the Comprehensive Geriatric Assessment and accepted as determinants of frailty. These frailty dimensions include cognitive status, general health status, functional independence, social support, medication use, nutrition, mood, continence and functional status. The scale consists of 11 items in total. The 'clock test' is used to assess cognitive status and the 'Timed Up and Go test' is used to assess functional performance.
Edmonton Frailty Scale | 3 months after the operation
  Edmonton Frailty Scale was developed by Rolfson et al. (2006) to assess frailty in elderly individuals. The scale consists of 9 frailty dimensions included in the Comprehensive Geriatric Assessment and accepted as determinants of frailty. These frailty dimensions include cognitive status, general health status, functional independence, social support, medication use, nutrition, mood, continence and functional status. The scale consists of 11 items in total. The 'clock test' is used to assess cognitive status and the 'Timed Up and Go test' is used to assess functional performance.
Causes of Kinesiophobia Scale | 3 days after the operation
  The Causes of Kinesiophobia Scale (CNS) is a 20-question questionnaire developed by Kocjan and Knapik (2015) to diagnose and determine the causes of motor inactivity. The CNS consists of a total of 20 questions and two subscales.
Causes of Kinesiophobia Scale | 3 weeks after the operation
  The Causes of Kinesiophobia Scale (CNS) is a 20-question questionnaire developed by Kocjan and Knapik (2015) to diagnose and determine the causes of motor inactivity. The CNS consists of a total of 20 questions and two subscales.
Causes of Kinesiophobia Scale | 3 months after the operation
  The Causes of Kinesiophobia Scale (CNS) is a 20-question questionnaire developed by Kocjan and Knapik (2015) to diagnose and determine the causes of motor inactivity. The CNS consists of a total of 20 questions and two subscales.
Care Dependency Scale | 3 days after the operation
  The Care Dependency Scale is a scale based on Virginia Henderson's human needs and developed to assess the care dependency status of patients. The Care Dependency Scale includes various physical and psychological aspects and provides a comprehensive assessment of the patient's care dependency. This scale was developed by Dijkstra in 1998. The items included in the scale are nutrition, continence, body posture, mobility, day/night cycle, dressing and undressing, body temperature, body cleanliness, avoiding hazards, communication, communicating with others, worshipping, following rules, daily activities, recreational activities and learning ability.
Care Dependency Scale | 3 weeks after the operation
  The Care Dependency Scale is a scale based on Virginia Henderson's human needs and developed to assess the care dependency status of patients. The Care Dependency Scale includes various physical and psychological aspects and provides a comprehensive assessment of the patient's care dependency. This scale was developed by Dijkstra in 1998. The items included in the scale are nutrition, continence, body posture, mobility, day/night cycle, dressing and undressing, body temperature, body cleanliness, avoiding hazards, communication, communicating with others, worshipping, following rules, daily activities, recreational activities and learning ability.
Care Dependency Scale | 3 months after the operation
  The Care Dependency Scale is a scale based on Virginia Henderson's human needs and developed to assess the care dependency status of patients. The Care Dependency Scale includes various physical and psychological aspects and provides a comprehensive assessment of the patient's care dependency. This scale was developed by Dijkstra in 1998. The items included in the scale are nutrition, continence, body posture, mobility, day/night cycle, dressing and undressing, body temperature, body cleanliness, avoiding hazards, communication, communicating with others, worshipping, following rules, daily activities, recreational activities and learning ability.

CONTACTS AND LOCATIONS:
Overall Officials: Halise Cinar, Principal Investigator — Aydin Adnan Menderes University, Turkey; Nurdan Gezer, Study Chair — Aydin Adnan Menderes University, Turkey
Locations (1):
- Aydin Adnan Menderes Üniversity, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No